CLINICAL TRIAL: NCT03625752
Title: Optimization of Non-Invasive Brain Stimulation for Diabetic Neuropathy
Brief Title: Optimization of NIBS for Diabetic Neuropathy Neuropathic Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Highland Instruments, Inc. (Industry)
Responsible Party: Principal Investigator, Ciro Ramos Estebanez, MD., Ph.D., Neurology faculty, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY20180314-2/20201584; NCT05469074 (obsolete NCT alias)
Record Dates: First submitted 2018-07-27; First posted 2018-08-10 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Neuropathies; Chronic Pain
MeSH Terms: conditions — Diabetic Neuropathies; Chronic Pain

STUDY DESIGN:
Intervention Model Description: single-center, double-blinded, placebo controlled, randomized study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Comparator: Active tDCS + Active TUS (Active Comparator): Subjects in the experimental group will undergo 20 minutes of active transcranial direct current stimulation (tDCS) and active transcranial ultrasound (TUS).
  Interventions: Device: Active Comparator: Active tDCS + Active TUS
- Sham (Sham Comparator): Subjects in the sham group will undergo 20 minutes of sham transcranial direct current stimulation (tDCS) and sham transcranial ultrasound (TUS).
  Interventions: Device: Sham

INTERVENTIONS:
Device: Active Comparator: Active tDCS + Active TUS — Device: transcranial Direct Current Stimulation (tDCS) Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2mA. The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes. Device: Transcranial Ultrasound (TUS) Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.
  Arms: Active Comparator: Active tDCS + Active TUS
Device: Sham — Device: SHAM Comparator Device: transcranial Direct Current Stimulation (tDCS) Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2mA. The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes. Device: Transcranial Ultrasound (TUS) Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.
  Arms: Sham

SUMMARY:
The purpose of this study is to assess the effects of Transcranial Direct Current Stimulation (tDCS) in combination with Transcranial ultrasound (TUS) for the treatment of pain and functional limitations in subjects with Diabetic Neuropathic Pain.

DETAILED DESCRIPTION:
Active stimulation will be compared with compared to SHAM stimulation in DNP patients.

20 DNP patients, 10 per group, receive stimulation or sham for 5 consecutive days, 20 min/day, followed by 2, 4, and 6 weeks post-therapy. 9 visits plus screening/baseline (total 10 visits).

Subsequently, 40 DNP patients will be enrolled, 20 per group, giving 5 consecutive days, 20 min/day, followed by 2 weeks of bi-weekly stimulation or sham for 20 min/day (total stimulations n=9) and follow-ups at 2, 4, 6, & 8 weeks post-stim): 13 visits plus screening/ baseline (total 14 visits).

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent to participate in the study.
2. Subjects between 40 to 80 years old.
3. Having diabetic neuropathic pain, involving at least 1 foot, with existing pain for at least 6 months, and having pain on at least half the days in the past 6 months with an average of at least a 4 on a 0-10 VAS scale).
4. Having pain resistant to common analgesics and medications for first-line therapy of chronic pain such as Tylenol, Aspirin, Ibuprofen, Soma, Parafon Forte DCS, Zanaflex, Codeine, etc.
5. Must have the ability to feel pain as self-reported.

Exclusion Criteria:

1. Subject is pregnant.
2. Contraindications to tDCS in conjunction with TUS, i.e. metallic implant in the brain or implanted brain medical devices
3. History of alcohol or drug abuse within the past 6 months as self-reported.
4. Use of carbamazepine within the past 6 months as self-reported.
5. Suffering from severe depression (with a PHQ 9 score of ≥ 10).
6. History of neurological disorders as self-reported.
7. History of unexplained fainting spells as self-reported.
8. History of severe head injury resulting in more than a momentary loss of consciousness as self-reported.
9. History of neurosurgery as self-reported.
10. Unstable pain (defined as pain intensities that vary by more than 4 points on 0-10 VAS scale over the 1-week period of trial run-in).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Changes in pain as measured by the Visual Analog Scale (VAS) | Measured for approximately 3 months
  The scale will assess a patient's pain intensity on a scale from 0 (no pain) to 10 (worst pain imaginable). Changes in VAS for Pain will be measured to determine whether anodal transcranial direct current stimulation (tDCS) in conjunction with transcranial ultrasound (TUS) (applied in a diagnostic mode) is effective in reducing pain of subjects with diabetic neuropathic pain.

SECONDARY OUTCOMES:
Changes in the Verbal Rating Scale (VRS) for Pain | Measured for approximately 3 months
  The VRS for Pain is a categorical scale of pain with categories: none, mild, moderate, severe pain intensity. Changes in VRS for Pain will be measured in order to determine whether anodal transcranial direct current stimulation (tDCS) in conjunction. with transcranial ultrasound (TUS) (applied in a diagnostic mode) is effective in reducing pain of subjects with diabetic neuropathic pain.
Changes in Conditional Pain Modulation | Measured for approximately 3 months
  Changes in Conditional Pain Modulation (CPM) will be measured in order to determine whether anodal transcranial direct current stimulation (tDCS) in conjunction with transcranial ultrasound (TUS) (applied in a diagnostic mode) is effective in increasing the pain pressure threshold in subjects with diabetic neuropathic pain.
Changes in Visual Analog Scalefor Mood (VAMS) | Measured for approximately 3 months
  The VAS for Mood will investigate Anxiety, Depression, Stress, and Sleepiness. The Subscales are as follows:
  The anxiety scale will assess a patient's anxiety on a scale from 0 (not anxious) to 10 (very anxious).
  The depression scale will assess a patient's depression on a scale from 0 (not depressed) to 10 (very depressed).
  The stress scale will assess a patient's stress on a scale from 0 (not stressed) to 10 (very stressed).
  The sleepiness scale will assess a patient's depression on a scale from 0 (not sleepy) to 10 (very sleepy).
Montreal Cognitive Assessment | Measured for approximately 3 months
  The investigators will monitor the safety of tDCS and TUS in subjects by measuring any changes in cognition. Scores range from lowest being 0 to highest being 30.
4-choice reaction time | Measured for approximately 3 months
  This is an attentional task that measures the time for a subject response to stimuli (in seconds) with shorter times being better.
N-back tests | Measured for approximately 3 months
  Assesses registration and immediate recall on a scale of the number of items correctly responded to
Electroencephalography | Measured for approximately 3 months
  Investigators will measure electroencephalogram (EEG) electrical activity (EEG amplitude and EEG frequency) as function of time.
Walking test | Measured for approximately 3 months
  The investigators will measure if there are changes in the walking speed, gait asymmetry, stride length, and walking smoothness of the subject from the beginning of the study to the end
Functional reach test | Measured for approximately 3 months
  The investigators will measure changes in subjects ability to complete the functional reach test across the duration of study.
Study 36-Item Short Form (SF-36) | Measured for approximately 3 months
  This is a health survey using a scale from 0 (worst) to 100 (best)
Patient Health Questionnaire (PHQ-9) | Measured for approximately 3 months
  This questionnaire screens for depression with a score of 0 (best) to 27 (worst)
American Pain Foundation Pain and Medication Diary | Measured for approximately 3 months
  The pain sub-scale measures pain intensity from 0 (best) to 10 (worst)
Multidimensional Pain Inventory (MPI) | Measured for approximately 3 months
  This pain scale measures aspects of pain from 0 (best) to 6 (worst)
Brief Pain Inventory-DPN | Measured for approximately 3 months
  This pain scale measures aspects of pain from 0 (no pain) to 10 (worst)
Adverse events | Measured for approximately 3 months
  At each session after stimulation begins, subjects will complete a questionnaire to evaluate potential adverse effects of stimulation (headache, neck pain, mood alterations, and seizures) on a 5-point scale (0 being best and 5 worst). The scale will also be administered at the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Salim Hayek, MD PhD, Principal Investigator — University Hospitals Cleveland Medical Center/ Case Western Reserve University
Locations (2):
- United States (2):
  - Ciro Ramos Estebanez, Chicago, Illinois
  - University Hospitals Cleveland Medical Center/ Dahms Clinical Research Unit, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No